CLINICAL TRIAL: NCT05784025
Title: Gait Training With antiGRAVIty TREadmill 'Alter-G', in Patients With ParkinSON Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Roberta Cellini, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GRAVITESON
Record Dates: First submitted 2023-03-14; First posted 2023-03-24 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AlterG (Experimental): Traditional rehabilitation program plus robotic rehabilitation making use of the antigravity AlterG device
  Interventions: Device: AlterG
- Control (No Intervention): Standard rehabilitation program

INTERVENTIONS:
Device: AlterG — Experimental device reducing weight perception by inducing a no-gravity environment which facilitates the execution of rehabilitation programs
  Arms: AlterG

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disease characterized mainly by motor symptoms, in particular rigidity, akinesia, tremor, which are associated with postural reflex deficits, impaired balance and gait deficit, with consequent significant limitation and impairment not only of functional independence but also of social and community life.

Postural instability leads to the appearance of accidental falls due: to the sudden loss of balance which is associated with the impossibility of implementing the right compensatory parachute reflexes; This can lead to serious consequences in these patients, in particular musculoskeletal trauma. In addition, progressive alterations of the gait lead to the phenomenon of freezing or freezing (FOG), in itself the cause of frequent falls. Physiotherapy in PD, including cueing techniques, treadmill training, and cognitive movement strategies, has been shown to improve balance and gait in PD patients. When we talk about subjects affected by PD. Often the painful symptomatology is an obstacle to intensive rehabilitation treatment.

The study conducted by José Fidel Baizabal-Carvallo (10-2020) showed that a training program that includes relatively low workloads provided benefits in different aspects of the Freezing of Gait and greater mobility, with a lower incidence of falls and consequently of musculo-articular damaging events.

The Alter-G M320 anti-gravity treadmill allows a lifting force to be applied evenly and comfortably to the patient's body. Lightening the body up to 80% of the weight, thanks to the pressure variation inside the air envelope, Alter-G allows patients or athletes to walk and run respecting motor patterns without compromising the biomechanics of eccentric movement. Through precise air pressure control (DAP - Differential Air Pressure) allows to improve aerobic conditioning activities without increasing the risk of stress injury. In addition, compared to traditional rehabilitation in the pool, AlterG allows maximum precision in the alleviation of discharge, being able to vary the load by one percentage point at a time.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disease characterized mainly by motor symptoms, in particular rigidity, akinesia, tremor, which are associated with postural reflex deficits, impaired balance and gait deficit, evident in particular in the onset phase and during the first years of the disease, which are associated in a more advanced stage cognitive and behavioral disorders, with consequent significant limitation and impairment not only of functional independence but also of social and community life. Although drug treatment has significantly modified the natural course of the disease, the gait and balance deficits worsen over time, leading progressively to higher levels of disability. In particular, postural instability leads to the appearance of accidental falls due: to the sudden loss of balance which is associated with the impossibility of implementing the right compensatory parachute reflexes; This can lead to serious consequences in these patients, in particular musculoskeletal trauma, including fractures of the femur, which can compromise not only the quoad valetudinem but also the quoad vitam. In addition, progressive alterations of the gait lead to the phenomenon of freezing or freezing (FOG), in itself the cause of frequent falls. Physiotherapy in PD, including cueing techniques, treadmill training, and cognitive movement strategies, has been shown to improve balance and gait in PD patients. When we talk about subjects affected by PD, with an average age generally over 65 years, we refer to a slice of the population defined as elderly. In the elderly patient all the physical and psychological problems inherent in the disease, starting with the pain phenomenon, acquire a particular significance in relation to the reduced performance status linked to age and other comorbidities, where chronic-degenerative diseases such as osteoarthritis and osteoporosis play a role of significant impact. Often the painful symptomatology is an obstacle to intensive rehabilitation treatment.

The study conducted by José Fidel Baizabal-Carvallo (10-2020) showed that a training program that includes relatively low workloads provided benefits in different aspects of the Freezing of Gait and greater mobility, with a lower incidence of falls and consequently of musculo-articular damaging events.

The Alter-G M320 anti-gravity treadmill, developed at NASA, allows a lifting force to be applied evenly and comfortably to the patient's body. Lightening the body up to 80% of the weight, thanks to the pressure variation inside the air envelope, Alter-G allows patients or athletes to walk and run respecting motor patterns without compromising the biomechanics of eccentric movement. This tool allows movement to elderly patients, the recovery of motor efficiency following surgery, learn to walk with joint or limb prostheses, carry out a real recovery in the neurological field, rehabilitate patients with injuries to the lower limbs, achieve effective aerobic conditioning, carry out specific conditioning programs. Through precise air pressure control (DAP - Differential Air Pressure) allows to improve aerobic conditioning activities without increasing the risk of stress injury. In addition, compared to traditional rehabilitation in the pool, AlterG allows maximum precision in the alleviation of discharge, being able to vary the load by one percentage point at a time.

More specifically, this technology allows:

* Recover stress fractures on bone structures subject to functional overload.
* Orthopedic rehabilitation before and after surgery
* Neurological rehabilitation for the recovery of gait control in patients affected by STROKE or comatose states as a result of severe brain injuries, Parkinson's disease, Multiple Sclerosis.
* Facilitate functional recovery of joints in patients undergoing reconstructive surgery in the lower limbs.
* Strengthening training of elderly patients
* Amateur and competitive sports preparation.
* Lose weight without damaging joints.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* Evidence of freezing of gait
* Age between 50 and 85
* Hoehn Yahr staging between II and III
* Mini Mental State Examination ≥ 24 (corrected for age and education)

Exclusion Criteria:

* Presence of musculoskeletal diseases
* Presence of severe visual and/or hearing impairment
* Presence of known heart or lung diseases contraindicating physical exercise
* Diagnosis of Parkinsonisms
* Presence of implanted cardiac pacemaker or programmable pump systems

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait performance | 12 months
  change in meters at the 6 minute walking test
Gait performance | 12 months
  change in minutes needed to perform the 10 meter walking test
risk of falls | 12 months
  incidence of fall episodes

SECONDARY OUTCOMES:
quality of life | 12 months
  changes in the EQ-5D (EuroQol five dimensions questionnaire) score
mood | 12 months
  changes in the Hamilton Anxiety Inventory score

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Cellini, Dr, Principal Investigator — IRCCS Centro Neurolesi Bonino Pulejo
Locations (1):
- Roberta Cellini, Messina, Italy

IPD SHARING:
Plan to Share IPD: No